CLINICAL TRIAL: NCT01635634
Title: Randomized Controlled Pilot Trial: The Effectiveness of Cupping in Patients With Fibromyalgia
Brief Title: Cupping in Fibromyalgia
Acronym: CuFib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr. med., Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CuFib
Record Dates: First submitted 2012-07-03; First posted 2012-07-09 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Cupping
MeSH Terms: conditions — Fibromyalgia | interventions — Cupping Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham Cupping (Sham Comparator): Dry Cupping Therapy 5 serial treatments twice weekly 4-8 cups at the upper and lower back
  Interventions: Other: Cupping therapy
- Cupping Therapy (Experimental): Dry Cupping 5 serial treatments twice weekly 4-8 cups at the upper and lower back
  Interventions: Other: Cupping therapy
- Wait list (No Intervention): Wait list control no specific intervention for 3 weeks study period

INTERVENTIONS:
Other: Cupping therapy — Cups are placed at the skin; local suction is created on the skin; it mobilizes blood flow; the suction is created by a mechanical device (Pneumatron, Pneumed, Germany)
  Arms: Cupping Therapy; Sham Cupping

SUMMARY:
The purpose of this randomized controlled study is to determine the effectiveness of cupping in patients with fibromyalgia compared to sham cupping.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* FMS diagnosis according to AWMF Guidelines,
* necessary documents: medical records
* Pain intensity > 45mm VAS
* Participation in cupping twice weekly on appointment

Exclusion Criteria:

* pregnancy
* other study participation
* pain due to other rheumatic disease
* major psychiatric disorder
* substance abuse
* severe somatic disorder (cancer)
* injections, acupuncture, neural therapy within the past 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Day 18
  Pain on a 100mm visual analog scale

SECONDARY OUTCOMES:
Pain Intensity | Day 200
  Pain intensity measured on a 100mm visual analog scale
Fatigue | Day 18
  Fatigue measured by the Multidimensional Fatigue Inventory (MFI) (Smets, Garssen, Bonke et al., 1995
Fatigue | Day 200
  Fatigue measured by the Multidimensional Fatigue Inventory (MFI) (Smets, Garssen, Bonke et al., 1995
Sleep Quality | Day 18
  measured by the Pittsburgh Sleep Quality Index (PSQI) (Buysse et al. 1989)
Sleep Quality | Day 200
  measured by the Pittsburgh Sleep Quality Index (PSQI) (Buysse et al. 1989)
Quality of life | Day 18
  measured by the SF-36 (Bullinger & Kirchberger, 1998)
Quality of life | Day 200
  measured by the SF-36 (Bullinger & Kirchberger, 1998)
Medication | Day 18
  measured by a medication log, daily entering of used drugs
adverse events | Day 18
  all adverse events
Pressure pain sensitivity | Day 18
  using an electronic algometer (Somedic, Sweden) to determine threshold of pain perception on predefined muscles
Disability | Day 18
  measured by the FI (fibromyalgia impact questionnaire) (Offenbaecher, Waltz, Schoeps , 2000)
Disability | Day 200
  measured by the FI (fibromyalgia impact questionnaire) (Offenbaecher, Waltz, Schoeps , 2000)

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, MD, Prof, Principal Investigator — University of Duisburg-Essen
Locations (1):
- Klinik für Naturheilkunde, Essen, Germany

REFERENCES:
- [Background] Lauche R, Spitzer J, Schwahn B, Ostermann T, Bernardy K, Cramer H, Dobos G, Langhorst J. Efficacy of cupping therapy in patients with the fibromyalgia syndrome-a randomised placebo controlled trial. Sci Rep. 2016 Nov 17;6:37316. doi: 10.1038/srep37316. PMID 27853272
- See also: Homepage of the Clinic — http://www.kliniken-essen-mitte.de/leistung/fachabteilungen/naturheilkunde-u-integrative-medizin/home.html